CLINICAL TRIAL: NCT01084577
Title: A Prospective, Multi-centre, Randomized, Open-label, Parallel, Comparative Study to Evaluate Effects of AQUACEL® Ag Dressing and Urgotul® Silver Dressing on Healing of Chronic Venous Leg Ulcers
Brief Title: AQUACEL® Ag Dressing and Urgotul® Silver Dressing on Healing of Chronic Venous Leg Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Dheerendra Kommala, MD, Convatec Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CW-0142-09-U354
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Leg Ulcer
MeSH Terms: conditions — Leg Ulcer

ARMS (2):
- Urgotul® Silver (Active Comparator): Urgotul® Silver for four weeks followed by Urgotul® for the remaining 4 weeks.
  Interventions: Device: Urgotul® Silver
- AQUACEL® Ag (Active Comparator): AQUACEL® Ag dressing for four weeks followed by AQUACEL® for the remaining 4 weeks.
  Interventions: Device: AQUACEL® Ag

INTERVENTIONS:
Device: AQUACEL® Ag — AQUACEL® Ag dressing for four weeks followed by AQUACEL® for the remaining 4 weeks.
  Arms: AQUACEL® Ag
Device: Urgotul® Silver — Urgotul® Silver for four weeks followed by Urgotul® for the remaining 4 weeks.
  Arms: Urgotul® Silver

SUMMARY:
A prospective, comparative, randomised study to compare the effects on ulcer healing of AQUACEL® Ag dressing when used for 4 weeks followed by treatment with AQUACEL® for 4 weeks to Urgotul® Silver dressing followed by Urgotul® for 4 weeks on subjects with venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years, willing and able to provide written informed consent.
* Subjects who have an ankle to brachial pressure index (ABPI) of 0.8 or greater.
* Subjects who have a venous leg ulcer (i.e. CEAP classification of C6), with duration less than 24 months and size ranging between 5 cm2-40 cm2 .
* Subjects' leg ulcers will meet at least 3 of the 5 following clinical signs: pain between 2 dressing changes, perilesional skin erythema, oedema, foul odour, and heavy exudation.
* Subjects agree to wear compression therapy daily in combination with the trial dressing.

Exclusion Criteria:

* Subjects with a history of skin sensitivity to any of the components of the study product.
* Subjects who have had current local or systemic antibiotics in the week prior to inclusion.
* Subjects whose leg ulcers are clinically infected or erysipelas, malignant, or who have had recent deep venous thrombosis or venous surgery within the last 3 months.
* Subjects who have a progressive neoplastic lesion treated by radiotherapy or chemotherapy, or on-going treatment with immunosuppressive agents or high dose corticosteroids.
* Subjects who have participated in a clinical study within the past 3 months.
* Subjects who are pregnant or breastfeeding (in accordance with the Urgotul® Silver package insert).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Wound area reduction from baseline (relative) | 8 weeks

SECONDARY OUTCOMES:
Wound closure | 8 weeks
Clinical evolution of the wound | 8 weeks
  presence of each of the 5 selected clinical signs
Tolerance | 8 weeks
  occurrence of local adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dheerendra Kommala, MD, Study Director — ConvaTec Inc.
Locations (56):
- Denmark (3):
  - Arhus Universitets Hospital (#47), Aarhus
  - Bispebjerg Universitets Hospital (#45), Copenhagen
  - Odense Universitets Hospital (#46), Odense
- France (8):
  - (#35), Paris, Neuilly Sur Siene
  - 37 Bd Bury (#42), Angoulême
  - CH de La Fere, (#44), La Fère
  - Clinique des Augustines (#38), Malestroit
  - 19 rue des Clers (#37), Metz
  - Hopital Brocca, 54/56 rue Pascal (#41), Paris
  - Centre de Sante (#36), Paris
  - Clinique Pasteur (#40), Toulouse
- Germany (4):
  - Praxis Dr Thinesse-Mallwitz (#31), München, Faustlestr 3
  - Hautarztpraxis Dr Klovekorn (#33), Gilching, Romerstr 4
  - Chirurgisches Zentrum Bethanien (#34), Frankfurt am Main, Usinger Str 5
  - Arztin fur Allgemeinmedizin (#30), München
- Poland (15):
  - Poradnia Medycyny Paliatywnej, Hospicjum Palium, SK im. Przemienienia Panskiego nr.1(#49), Poznan, Os. Rusa 25a
  - NZoZ SEP-MED (#59), Warsaw, Ul. Hoza 19
  - Centr. Med. Beluga-Med, NZOZ (#53), Krakow, Ul. Obopolna 4a
  - Poradnia Chorob MIKOMED (#55), Lodz, Ul. Plugowa 51/53
  - NZOZ Por. Chrurgiczna (#52), Strzelce Opolskie, Ul. Powstancow Slaskich 9
  - Centr. Diagnostyki Ginek.-Poloz. (#51), Opole, Ul.1-go Maja 9/69-73
  - Szpital Woj.w Bielsku-Bialej (#61), Bielsko-Biala, ul.Armii Krajowej 101
  - Poradnia Chirurgiczna Szpital, Specjalistyczny nr.2 (#50), Bytom, ul.Batorego 15
  - Nzoz Certus (#64), Lodz, ul.Kopernika 67-69
  - Venavita (#63), Poznan, ul.Kurpiowska 8/5
  - Specjal.Pomoc Med.MEDSERVICE (#56), Zabrze, ul.M.Sklodowskiej-Curie 34
  - SPZOZ nr.1 Przyszpitalna Por. (#58), Rzeszów, ul.Rycerska 4
  - Nzoz Serce Sercu (#62), Mogilany, ul.Sw.Bartlomieja Apostola 21
  - CF Centrum Flebologii (#60), Warsaw, ul.Witosynskiego 5
  - SPZOZ UM w Lodzi (#54), Ul. Narutowicza 96, Łódź Voivodeship
- United Kingdom (26):
  - Vestry Close Health Clinic (#8), Luton, Bedfordshire
  - Chalfont and Gerrards Cross Hospital (#14), Chalfont Saint Peter, Buckinghamshire
  - Wound Healing Research Unit (#1), Heathpark, Cardiff
  - University Hopital (#15), West Midlands, Coventry
  - Hainult Health Centre (#24), Chigwell, Essex
  - Rayleigh Clinic (#19), Rayleigh, Essex
  - Southend University Hopital (#20), Westcliff-on-Sea, Essex
  - Distric Nurses, The Wilson Practice, Alton Health Centre (#9), Alton, Hampshire
  - Fareham College Specialist Leg Care Centre (#13), Fareham, Hampshire
  - Southampton Hospital (#6), Southampton, Hampshire
  - St Mary's Hospital (#7), Armley, Leeds
  - Forest Primary Care Center (#18), Edmonton, London
  - Tissue Viability Service NHS Harrow PCT (#26), Harrow, Middlesex
  - Norwich Community Hospital (#21), Norwich, Norfolk
  - Tissue Viability Service, The Willows, Centre for Health Care (#11), Weaste, Salford
  - Mayday University Hospital Wound Clinic (#10), Thornton Health, Surrey
  - Goldsworth Park Health Centre (022), Woking, Surrey
  - Neath Port Talbot Hospital (#17), Port Talbot, West Glamorgan
  - City Hospital (#12), Birmingham, West Midlands
  - University Hospital (#15), Coventry, West Midlands
  - Cross Street Health Centre (#4), Dudley, West Midlands
  - Solihull Hospital (#5), Solihull, West Midlands
  - Arrowe Park Hospital (#2), Upton, Wirral
  - Tissue Viability Consultancy (#3), Eastbourne
  - Royal Free Hospital (#23), London
  - Stourport Health Centre (#16), Worcestershire